CLINICAL TRIAL: NCT07191626
Title: Pulsed Field Ablation of Superior Vena Cava in Addition to Pulmonary Vein in Paroxysmal Atrial Fibrillation: A Multicenter Randomized Controlled Trial (PASPA Study)
Brief Title: Pulsed Field Ablation of SVC and PV in Paroxysmal Atrial Fibrillation (PASPA Study)
Acronym: PASPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PASPA-2025-001
Record Dates: First submitted 2025-09-08; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Paroxysmal Atrial Fibrillation; Paroxysmal Atrial Fibrillation (PAF)
Keywords: Paroxysmal, Catheter Ablation; Catheter Ablation; Pulsed Field Ablation; Pulmonary Vein Isolation; Superior Vena Cava Isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design. Eligible participants are randomly assigned in a 1:1 ratio to one of two study arms: (1) pulsed field ablation guided pulmonary vein isolation (PVI alone), or (2) pulsed field ablation guided pulmonary vein isolation plus superior vena cava isolation (PVI + SVC). Each participant receives only the intervention of the assigned arm. Randomization is stratified by study center to ensure balanced allocation across all 20 participating centers.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI + SVCI (Experimental): Catheter ablation procedure using a Pulsed Field Ablation system to achieve electrical isolation of all pulmonary veins AND the superior vena cava.
  Interventions: Procedure: PFA - PV + SVCI
- PVI only (Active Comparator): Catheter ablation procedure using a Pulsed Field Ablation system to achieve electrical isolation of all four pulmonary veins ONLY.
  Interventions: Procedure: PFA - PVI only

INTERVENTIONS:
Procedure: PFA - PV + SVCI — Catheter ablation procedure using a Pulsed Field Ablation system to achieve electrical isolation of all four pulmonary veins AND the superior vena cava.
  Arms: PVI + SVCI
Procedure: PFA - PVI only — Catheter ablation procedure using a Pulsed Field Ablation system to achieve electrical isolation of all four pulmonary veins only. No ablation is performed in the superior vena cava.
  Arms: PVI only

SUMMARY:
The PASPA study is a multicenter, randomized trial comparing Pulmonary Vein Isolation (PVI) alone versus PVI plus Superior Vena Cava Isolation (SVCI) using Pulsed Field Ablation (PFA) in patients with paroxysmal atrial fibrillation (PAF).

650 participants will be followed for 12 months. The main goal is to see if adding SVCI reduces arrhythmia recurrence without increasing complications such as phrenic nerve injury or sinus node dysfunction.

DETAILED DESCRIPTION:
The PASPA study addresses the limitations of traditional pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (PAF), where recurrence rates remain significant due to non-pulmonary vein triggers such as the superior vena cava (SVC). Traditional ablation near the SVC carries risks of phrenic nerve and sinus node injury, and acute isolation success rates are only 75%-85%. Pulsed Field Ablation (PFA) selectively ablates cardiomyocytes through irreversible electroporation while sparing adjacent nerves and vessels, allowing safer SVC isolation. This prospective, multicenter, randomized controlled trial will enroll 650 patients with documented PAF, randomly assigned to PVI alone or PVI plus SVC isolation (SVCI) using PFA. Participants will be followed for 12 months with 7-day Holter monitoring at 3, 6, and 12 months. The primary endpoint is freedom from atrial fibrillation, atrial flutter, or atrial tachycardia episodes ≥30 seconds at 12 months. Secondary endpoints include atrial fibrillation burden and procedure-related complications such as phrenic nerve injury, cardiac tamponade, and sinus node dysfunction. Preliminary animal and pilot human studies indicate that PFA achieves 100% acute SVC isolation with minimal complications. The study aims to determine whether adding SVCI to PVI improves efficacy in PAF without increasing procedural risks, providing evidence to guide standardized ablation strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Documented paroxysmal AF (episodes self-terminating within 7 days), evidenced by ECG, Holter, or event monitor
2. Age between 18 and 80 years
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Intracardiac thrombus (left atrium or left atrial appendage)
2. Left atrial anterior-posterior diameter > 60 mm
3. Absolute contraindication to anticoagulation therapy
4. Stroke or myocardial infarction within 1 month prior to enrollment
5. Uncontrolled hyperthyroidism
6. Pregnancy or planning pregnancy
7. Life expectancy less than 1 year
8. Previous atrial fibrillation ablation procedure
9. Known or suspected AF triggers primarily originating from the SVC (based on pre-procedure mapping, if available)
10. Inability or unwillingness to participate in the study or comply with follow-up requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia recurrence at 12 Months | 12 month
  Proportion of participants without recurrence of atrial fibrillation, atrial flutter, or atrial tachycardia lasting ≥30 seconds, as assessed by 7-day continuous ambulatory ECG monitoring, during the 12-month follow-up period after ablation.

SECONDARY OUTCOMES:
Atrial Fibrillation Burden | 12 month
  The percentage of time spent in atrial fibrillation during the 7-day Holter monitoring periods, calculated as (total AF duration / total recording duration) * 100%.

OTHER OUTCOMES:
Composite Rate of Major Complications | 12 months
  The percentage of participants experiencing any of the major complications during the 12-month follow-up period.Major complications including phrenic nerve injury/palsy, cardiac tamponade, pericardial effusion requiring intervention, symptomatic sinus node dysfunction requiring pacemaker implantation, stroke/TIA, vascular access complications, and death.

CONTACTS AND LOCATIONS:
Overall Officials: zhifu guo, MD, Principal Investigator — The First Affiliated Hospital of Naval Medical University (Shanghai Changhai Hospital)
Locations (1):
- The First Affiliated Hospital of Naval Medical University (Shanghai Changhai Hospital). No. 168, Changhai Road, Yangpu District, Shanghai, China., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying the results will be shared after publication of the primary results, upon reasonable request and subject to approval by the study steering committee and applicable ethical/regulatory requirements.
Supporting Information: Study Protocol
Time Frame: Available starting 12 months after publication of the primary results, for a duration of 12 months.
Access Criteria: Access granted only to qualified researchers upon reasonable request. Only de-identified participant-level data will be shared. Requests are subject to sponsor approval.